CLINICAL TRIAL: NCT03879031
Title: Evaluation of the Responsiveness of the Bridge Tests in Subjects With Non-specific Subacute or Chronic Low Back Pain
Brief Title: Responsiveness of the Bridge Tests in Non-specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Paolo Pillastrini, Full professor - Director of the Masters in Musculoskeletal Physiotherapy - University of Bologna, University of Bologna
Other Study IDs: 1/Bridge
Record Dates: First submitted 2019-03-08; First posted 2019-03-18 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Low Back Pain
Keywords: lumbar; physical endurance; pain; disability; assessment
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients with low back pain: All outpatients with non-specific subacute or chronic low back pain will be submitted to a physical therapy program including:
  * information on pain mechanisms and the favorable nature of non-specific low back pain;
  * advice on positions, movements and activities recommended or advised against in people with low back pain, both at work and during leisure time;
  * active postural correction exercises, overactive muscles lengthening and weak musculature strengthening;
  * passive manual techniques, aimed at muscle relaxation and recovery of lumbar joint mobility.
  A cluster of Clinical tests to measure lumbar stability will be administrated before the starting of the first session and at the ending of the last session of the physical therapy program.
  Interventions: Diagnostic Test: Cluster of Clinical tests to measure lumbar stability

INTERVENTIONS:
Diagnostic Test: Cluster of Clinical tests to measure lumbar stability — All subjects will be submitted to a cluster of clinical test before the starting of the first session, and at the ending of the last session of the physical therapy program. This cluster will include:
  * Aberrant Movements (AM) Test,
  * Active Straight Leg Raise Test (ASLR) Test,
  * Supine Bridge Test (SuBT),
  * Right Side Bridge Test (RBT),
  * Left Side Bridge Test (LBT),
  * Prone Bridge Test (PrBT),
  * Passive Lumbar Extension (PLE) Test,
  * Prone Instability Test (PIT).

SUMMARY:
This observational study aims to investigate the internal responsiveness and external responsiveness of the Bridge Tests (supine bridge test, prone bridge test, and side bridge test) in relation to pain and disability, in subjects with subacute and chronic non-specific low back pain submitted to a physical therapy program.

DETAILED DESCRIPTION:
Time 0 (first session of the physical therapy treatment program)

The physical therapist will explain to each patient the purpose of the study and request informed consent and data processing consent. In the informed consent form will be specified that the study will concern some diagnostic tests and the study protocol will not influence the physical therapy treatment strategy in any way. Only those who give their consent will be included in the study and will fill in a booklet containing:

* socio-demographical, anthropometric and pain data;
* the Italian version of the Oswestry Disability Index (ODI-I);
* the Italian version of the 0-100 Numerical Rating Scale (NRS). Once completed, the questionnaires will be placed in a sealed envelope and delivered to the examiner.

The physical therapist will perform the following tests, without being aware of the results collected during the initial clinical evaluation and will record the tests results on a pre-printed sheet, which will then be inserted in the same envelope as well.

The tests performed are (in order of execution):

* Aberrant Movements (AM) Test,
* Active Straight Leg Raise (ASLR) Test,
* Supine Bridge Test (SuBT),
* Right Side Bridge Test (RBT),
* Left Side Bridge Test (LBT),
* Prone Bridge Test (PrBT),
* Passive Lumbar Extension (PLE) Test,
* Prone Instability Test (PIT).

The envelope containing the patient's data and the results of the tests will be sent to an independent subject, who will take care of the data collection and their insertion into the electronic database, assigning to each patient a numerical code as the only identification element.

The patients will be submitted to a physical therapy treatment for eight 30-minutes sessions, once a week.

Time 1 (at the end of the last session of the physical therapy treatment)

Those who have completed the physical therapy treatment will receive a final booklet containing the Italian version of the Oswestry Disability Index (ODI-I), the Numerical Rating Scale (NRS) and the Global Perceived Effect (GPE) Questionnaire. Once completed, these questionnaires will be placed in a sealed envelope and delivered to the examiner.

Without being aware of the outcome of the questionnaires contained in the final booklet, the same tests will be repeated:

* Aberrant Movements (AM) Test,
* Active Straight Leg Raise (ASLR) Test,
* Supine Bridge Test (SuBT),
* Right Side Bridge Test (RBT),
* Left Side Bridge Test (LBT),
* Prone Bridge Test (PrBT),
* Passive Lumbar Extension (PLE) Test,
* Prone Instability Test (PIT).

Test results will be recorded on a pre-printed sheet, which will then be inserted in the same envelope and send to the independent subject who is responsible for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific subacute or chronic low back pain (low back pain from 1 month or more, not related to specific pathologies);
* Low back pain, with or without irradiation to the lower limb, noted as ≥2 on a scale of 0-10;
* Good comprehension of written and spoken Italian Language;
* Informed consent.

Exclusion Criteria:

* Acute low back pain;
* Specific causes of low back pain (truma, herniated disc, vertebral deformity, fractures, dislocations);
* Central or peripheral neurologic signs;
* Systemic pathologies;
* Rheumatic disorders;
* Neuromuscular pathologies;
* Tumors;
* Cognitive deficits;
* Surgical interventions in the last six months prior to the study;
* Osteoporosis.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All outpatients entering the conservative physical therapy treatment for subacute or chronic non-specific low back pain in a Occupational Medicine Unit are considered eligible.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in low back pain over time | Time zero: at baseline - Time one: at the end of the last session of physical therapy treatment (8 weeks after Time zero)
  0-100 Numerical Rating Scale (NRS) for low back pain. This scale is arranged to measure the amount of perceived lumbar pain, from 0 (= no pain) to 100 (=maximum pain).
Changes in lumbar disability over time | Time zero: at baseline - Time one: at the end of the last session of physical therapy treatment (8 weeks after Time zero)
  Oswestry Disability Index - Italian version (ODI-I). This questionnaire measures disability related to low back pain in 10 different domains (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, and Traveling). The patients are asked to identify which of six statements in each domain applies to them at the time of evaluation. The sentences are arranged from no impairment (0) to maximum impairment (5). The scores for each domain are added together (range from 0 to 50) and multiplied by 2 which yields a Disability Index Score percent. If not all items are completed, the score is prorated by averaging the items completed and then multiplying it by 10. A Disability Index Score of 0% to 20% corresponds to minimal disability, 21% to 40% to moderate disability, 41% to 60% to severe disability, 61% to 80% crippled, and 81% to 100% indicates a patient that is either bed-bound or exaggerating their symptoms.

SECONDARY OUTCOMES:
Changes in Global Perceived Effect (GPS) questionnaire (Italian version) over time | At the end of the last session of physical therapy treatment (8 weeks after Time zero)
  The GPE is composed of one question on a 7-point Likert-type scale, evaluating the subjective self-reported improvement or deterioration after the intervention, from "fully improved" (score 1) to "fully worsened" (score 7). More specificaly, 1=fully improved; 2=much improved; 3=a little improved; 4=no change; 5= a little deterioration; 6=much deterioration; 7=fully worsened. GPE is widely used in the physical therapy literature.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, PT, Principal Investigator — University of Bologna
Locations (1):
- Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott JH, McCane B, Herbison P, Moginie G, Chapple C, Hogarty T. Lumbar segmental instability: a criterion-related validity study of manual therapy assessment. BMC Musculoskelet Disord. 2005 Nov 7;6:56. doi: 10.1186/1471-2474-6-56. PMID 16274487
- [Background] Alqarni AM, Schneiders AG, Hendrick PA. Clinical tests to diagnose lumbar segmental instability: a systematic review. J Orthop Sports Phys Ther. 2011 Mar;41(3):130-40. doi: 10.2519/jospt.2011.3457. Epub 2011 Feb 2. PMID 21289452
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Durall CJ, Greene PF, Kernozek TW. A comparison of two isometric tests of trunk flexor endurance. J Strength Cond Res. 2012 Jul;26(7):1939-44. doi: 10.1519/JSC.0b013e318237ea1c. PMID 22728944
- [Background] Ferrari S, Manni T, Bonetti F, Villafane JH, Vanti C. A literature review of clinical tests for lumbar instability in low back pain: validity and applicability in clinical practice. Chiropr Man Therap. 2015 Apr 8;23:14. doi: 10.1186/s12998-015-0058-7. eCollection 2015. PMID 25866618
- [Background] Fritz JM, Whitman JM, Childs JD. Lumbar spine segmental mobility assessment: an examination of validity for determining intervention strategies in patients with low back pain. Arch Phys Med Rehabil. 2005 Sep;86(9):1745-52. doi: 10.1016/j.apmr.2005.03.028. PMID 16181937
- [Background] Frymoyer JW, Selby DK. Segmental instability. Rationale for treatment. Spine (Phila Pa 1976). 1985 Apr;10(3):280-6. doi: 10.1097/00007632-198504000-00017. PMID 3992349
- [Background] Habets B, van Cingel RE, Ostelo RW. Reproducibility of a battery of commonly used clinical tests to evaluate lumbopelvic motor control. Phys Ther Sport. 2015 Nov;16(4):331-9. doi: 10.1016/j.ptsp.2015.02.004. Epub 2015 Mar 7. PMID 26254503
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Kasai Y, Morishita K, Kawakita E, Kondo T, Uchida A. A new evaluation method for lumbar spinal instability: passive lumbar extension test. Phys Ther. 2006 Dec;86(12):1661-7. doi: 10.2522/ptj.20050281. Epub 2006 Oct 10. PMID 17033040
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Mens JM, Huis In 't Veld YH, Pool-Goudzwaard A. The Active Straight Leg Raise test in lumbopelvic pain during pregnancy. Man Ther. 2012 Aug;17(4):364-8. doi: 10.1016/j.math.2012.01.007. Epub 2012 Feb 22. PMID 22365484
- [Background] Ozcan Kahraman B, Salik Sengul Y, Kahraman T, Kalemci O. Developing a Reliable Core Stability Assessment Battery for Patients with Nonspecific Low Back Pain. Spine (Phila Pa 1976). 2016 Jul 15;41(14):E844-E850. doi: 10.1097/BRS.0000000000001403. PMID 26679886
- [Background] Rabin A, Shashua A, Pizem K, Dar G. The interrater reliability of physical examination tests that may predict the outcome or suggest the need for lumbar stabilization exercises. J Orthop Sports Phys Ther. 2013 Feb;43(2):83-90. doi: 10.2519/jospt.2013.4310. Epub 2013 Jan 14. PMID 23321848
- [Background] Schellenberg KL, Lang JM, Chan KM, Burnham RS. A clinical tool for office assessment of lumbar spine stabilization endurance: prone and supine bridge maneuvers. Am J Phys Med Rehabil. 2007 May;86(5):380-386. doi: 10.1097/PHM.0b013e318032156a. PMID 17303961
- [Background] Stuge B, Veierod MB, Laerum E, Vollestad N. The efficacy of a treatment program focusing on specific stabilizing exercises for pelvic girdle pain after pregnancy: a two-year follow-up of a randomized clinical trial. Spine (Phila Pa 1976). 2004 May 15;29(10):E197-203. doi: 10.1097/00007632-200405150-00021. PMID 15131454
- [Background] Vanti C, Conti C, Faresin F, Ferrari S, Piccarreta R. The Relationship Between Clinical Instability and Endurance Tests, Pain, and Disability in Nonspecific Low Back Pain. J Manipulative Physiol Ther. 2016 Jun;39(5):359-368. doi: 10.1016/j.jmpt.2016.04.003. Epub 2016 May 7. PMID 27167368
- [Background] Vanti C, Ferrari S, Berjano P, Villafane JH, Monticone M. Responsiveness of the bridge maneuvers in subjects with symptomatic lumbar spondylolisthesis: A prospective cohort study. Physiother Res Int. 2017 Oct;22(4). doi: 10.1002/pri.1682. Epub 2017 Jan 6. PMID 28060461
- [Background] Weir A, Darby J, Inklaar H, Koes B, Bakker E, Tol JL. Core stability: inter- and intraobserver reliability of 6 clinical tests. Clin J Sport Med. 2010 Jan;20(1):34-8. doi: 10.1097/JSM.0b013e3181cae924. PMID 20051732